CLINICAL TRIAL: NCT06084650
Title: OCT and OCTA Deep Learning in Waldenström's Macroglobulinemia Patients
Brief Title: Optical Coherence Tomography (OCT) and OCT Angiography(OCTA) Deep Learning in Waldenström's Macroglobulinemia Patients
Acronym: OCTA
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, professor, Federico II University
Other Study IDs: 05809851
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- waldenstrom macroglobulinemia patients
- healthy patients matched age and sex without waldenstrom macroglobulinemia and ocular disease

SUMMARY:
This study evaluates the ability of deep learning to improve the knowledge about structural and vascular retinal changes in Waldenström's Macroglobulinemia patients, using optical coherence tomography angiography.

DETAILED DESCRIPTION:
Waldenstrom macroglobulinemia (mak-roe-glob-u-lih-NEE-me-uh) is a rare type of cancer that begins in the white blood cells.

The optical coherence tomography angiography represents a novel and noninvasive diagnostic technique that allows a detailed and quantitative analysis of retinal and choriocapillary vascular features. The study evaluates the changes in optical coherence tomography angiography features in Waldenstrom macroglobulinemia, elaborating these data with artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years

  * diagnosis of Waldenstrom Macroglobulinemia
  * absence of previous ocular surgery and congenital eye diseases.
  * absence of errors of refraction
  * absence of lens opacities
  * absence of low-quality OCT and OCTA images

Exclusion Criteria:

* • age younger than 18 years

  * previous ocular surgery and congenital eye diseases
  * errors of refraction
  * lens opacities
  * low-quality OCT and OCTA images

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participans were older than 18 years with diagnosis of Waldenstrom Macroglobulinemia. They did not present other ophthalmological disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
The measurements of retinal and choriocapillary vessel density in Waldenstrom Macroglobulinemia patients. | up to three months
  The parameters analyzed by optical coherence tomography angiography were: retinal and choriocapillary vessel density matched with clinical parameters resulted from the artificial pancreas device

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II" Naples, Italy, 80100 Contact: Gilda Cennamo, MD 00390817143731 xgilda@hotmail.com, Napoli, Italy